CLINICAL TRIAL: NCT02350608
Title: Pulse Waveform and ECG Analysis in Postoperative Cardiac Surgical Patients
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kati Järvelä, MD, PhD, Head of Cardiac Intensive Care Unit, Tampere University Hospital
Other Study IDs: R14013
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Blood Pressure; Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Noninvasive monitor — A novel technique on noninvasive blood pressure monitoring.

SUMMARY:
Observational study of 20 postoperative cardiac surgery patients. On admission to the ICU the patients will receive a noninvasive monitor recording arterial pulse waveform and ECG. The monitoring will continue to the ward for two days. The data will be compared with the routine monitoring methods.

DETAILED DESCRIPTION:
Observational study of 20 adult postoperative cardiac surgery patients. The observation will last from 0 to 2. postoperative day. On admission to the ICU the patients will receive a noninvasive monitor recording arterial pulse waveform and ECG. The monitoring will continue to the ward for two days. The data will be compared with the routine monitoring methods in the ICU and the ward.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patients, informed consent

Exclusion Criteria:

* Poor co-operation, age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Detection of arrythmia | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Jari Laurikka, Prof, Study Director — Tampere UH
Locations (1):
- Tampere University Hospital Heart Center, Tampere, Finland